CLINICAL TRIAL: NCT04239703
Title: Trifecta-Kidney cfDNA-MMDx Study: Comparing the DD-cfDNA Test to MMDx Microarray Test, Central HLA Antibody Test, and Histology.
Brief Title: Trifecta-Kidney cfDNA-MMDx Study
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Natera, Inc. (Industry); One Lambda (Unknown)
Responsible Party: Principal Investigator, Philip Halloran, Distinguished Professor, University of Alberta
Other Study IDs: ATAGC05
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant Rejection
Keywords: donor derived cell-free DNA; blood; kidney biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA isolated from kidney biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant biopsies for cause: The study population includes patients with a functioning kidney transplant undergoing a biopsy for clinical indications as standard of care.
  Interventions: Diagnostic Test: MMDx; Diagnostic Test: Prospera; Diagnostic Test: HLA antibody

INTERVENTIONS:
Diagnostic Test: MMDx — Portion of kidney transplant indication biopsy
Diagnostic Test: Prospera — Transplant patient blood sample
  Other Names: transplant patient blood sample
Diagnostic Test: HLA antibody — Transplant patient blood sample
  Other Names: transplant patient blood sample

SUMMARY:
Demonstrate the relationship between DD-cfDNA levels and HLA antibodies in blood, and the Molecular Microscope® (MMDx) Diagnostic System results in indication biopsies.

DETAILED DESCRIPTION:
There is a need for better screening of kidney transplant patients for rejection. Patients with kidney transplants are routinely tested (creatinine, urine protein, histology and donor specific antibody (DSA) as standard of care to detect rejection, but these tests are not adequate. Rejection is often missed by these tests (false negatives) and other processes such as acute kidney injury can produce false-positive results. Moreover, histology has a high interobserver disagreement diagnosing rejection, and cannot accurately assess acute injury. A definitive molecular assessment of rejection and injury in kidney biopsies has emerged - the Molecular Microscope® Diagnostic System (MMDx) - developed by the Alberta Transplant Applied Genomics Centre, University of Alberta. Now a new screening test is being introduced: the monitoring of donor-derived cell-free DNA (DD-cfDNA) released in the blood by the kidney during rejection. The Natera Inc DD-cfDNA Prospera® test is based on the massively multiplex PCR that targets 13,392 single nucleotide polymorphisms and targeted sequences are quantified by Next Generation Sequencing. The Prospera® test done on kidney transplant recipients detected "active rejection" and differentiated it from borderline rejection and no rejection. It is likely, however, that DD-cfDNA test may miss some T cell-mediated rejection (TCMR) cases and the distinction between early and fully developed antibody-mediated rejection (ABMR) was not tested. No study has actually examined the DD-cfDNA results in kidney transplants with acute or chronic kidney disease (AKI and CKD). DD-cfDNA measurements have only been correlated with histology, a flawed standard. DD-cf-DNA test must now be calibrated against MMDx that is based on global gene expression, the new standard for biopsy interpretation. The present study will calibrate centrally measured (Natera Inc) DD-cfDNA levels obtained at the time of an indication biopsy against the MMDx measurements of TCMR, and ABMR (early-stage, fully-developed, and late-stage), AK, and atrophy-fibrosis. We will compare blood DD-cfDNA measurements in 600 samples at the time of 300 indication biopsies to the MMDx results, as well as central assessment of HLA antibody (One Lambda) in 300 blood samples, interpreted centrally as DSA based on the tissue typing results. This study is an extension of the INTERCOMEX ClinicalTrials.gov Identifier: NCT01299168. We have collected 1203 kidney biopsies and 2422 corresponding blood samples. We extend this study to the total of 1400 biopsies and 2800 blood samples.

ELIGIBILITY:
Inclusion Criteria:

* All kidney transplant recipients undergoing a kidney biopsy for clinical indications, as determined by their physician or surgeon, will be eligible to enroll in the study.

Exclusion Criteria:

* Patients will be excluded from the study if they decline participation or are unable to give informed consent or multiple organ recipients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients with a functioning kidney transplant undergoing a biopsy for clinical indications as standard of care to determine the cause of their graft dysfunction (deterioration in graft function, delayed graft function, proteinuria).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Calibration of Prospera test for T cell-mediated rejection | 18 months
  Calibration of DD-cfDNA test cut-off values against the probability of T cell-mediated rejection in the biopsy as reported by MMDx.
Calibration of Prospera test for antibody-mediated rejection | 18 months
  Calibration of DD-cfDNA test cut-off values against the probability of antibody-mediated rejection in the biopsy as reported by MMDx.
Calibration of Prospera test for kidney injury | 18 months
  Calibration of DD-cfDNA test cut-off values against the probability of acute and chronic kidney injury in the biopsy as reported by MMDx.
Report calibrated Prospera test results for rejection | 6 months
  Report new DD-cfDNA test cut-off values for rejection
Report calibrated Prospera test results for kidney injury | 6 month
  Report new DD-cfDNA test cut-off values for acute and chronic kidney injury

SECONDARY OUTCOMES:
Determine if Prospera blood test can replace kidney biopsy test | 6 months
  Determine if Prospera test, as calibrated by this DD-cfDNA-HLA-MMDx study, will avoid need for indication biopsy when kidney transplant function deteriorates. This will be based on the consensus between participating clinicians.
Assessment of donor-specific antibody status | 6 months
  Report and compare the DSA status based on centralized and local HLA antibody measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD, PhD, Principal Investigator — University of Alberta
Locations (31):
- United States (11):
  - Tampa General Hospital, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - The Johns Hopkins University, School of Medicine, Baltimore, Maryland
  - Detroit Medical Center, Harper University Hospital of Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Barnes-Jewish Hospital, Washington University at St. Louis, St Louis, Missouri
  - University Hospitals Cleveland Medical Ctr., Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Intermountain Transplant Services, Murray, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Division of Nephrology & UW Organ Transplant Center University of Washington, Seattle, Washington
- Department of Nephrology, The Royal Melbourne Hospital 1 South East, Melbourne, Australia
- Canada (2):
  - University of Alberta, Department of Medicine, Edmonton, Alberta
  - ST. Paul's Hospital, 6A Providence Building, 1081 Burrard Street, Vancouver, British Columbia
- University Hospital Merkur Renal Division, Zagreb, Croatia
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Charite-Medical University of Berlin Department of Nephrology, Berlin, Germany
- Centre of Nephrology, Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Poland (11):
  - Department of Nephrology and Transplantation Medical University in Bialystok, Bialystok
  - University Hospital nr1 Bydgoszcz, Klinika Transplantologii, Bydgoszcz
  - Medical University of Gdańsk Klinika Nefrologii Transplantologii i Chorób Wewnętrznych, Gdansk
  - Medical University of Silesia, Katowice
  - Department of Transplantation and General Surgery, Wojewodzki Hospital, Poznan
  - Department of Nephrology, Transplantation and Internal Medicine, University Hospital n.2, Szczecin
  - Pomeranian Medical University, Samodzielny Publiczny Woj. Szpital Zespolony, Oddzial Nefrologii i Transplantacji Nerek, Szczecin
  - Medical University of Warsaw, Department of Transplantation Medicine, Nephrology and Internal Diseases, Warsaw
  - Transplant Medicine & Nephrology Clinic, Medical University of Warsaw, Warsaw
  - The Children's Memorial Health Institute, Department of Nephrology, Kidney Transplantation and Hypertension, Warsaw
  - Wroclaw Medical University, Department of Nephrology and Transplantation Medicine, Wroclaw
- Department of Nephrology, University Medical Centre, Ljubljana, Slovenia
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Background] Halloran PF, Madill-Thomsen KS. Donor-derived Cell-free DNA: A Step Forward in the Quest for Transplant Truth. Transplantation. 2025 Jun 1;109(6):910-914. doi: 10.1097/TP.0000000000005332. Epub 2025 Jan 28. No abstract available. PMID 39883025
- [Result] Halloran PF, Reeve J, Madill-Thomsen KS, Demko Z, Prewett A, Billings P; Trifecta Investigators. The Trifecta Study: Comparing Plasma Levels of Donor-derived Cell-Free DNA with the Molecular Phenotype of Kidney Transplant Biopsies. J Am Soc Nephrol. 2022 Feb;33(2):387-400. doi: 10.1681/ASN.2021091191. Epub 2022 Jan 20. PMID 35058354
- [Result] Halloran PF, Reeve J, Madill-Thomsen KS, Demko Z, Prewett A, Gauthier P, Billings P, Lawrence C, Lowe D, Hidalgo LG; the Trifecta Investigators. Antibody-mediated Rejection Without Detectable Donor-specific Antibody Releases Donor-derived Cell-free DNA: Results From the Trifecta Study. Transplantation. 2023 Mar 1;107(3):709-719. doi: 10.1097/TP.0000000000004324. Epub 2023 Feb 21. PMID 36190186
- [Result] Halloran PF, Madill-Thomsen KS, Reeve J. The Molecular Phenotype of Kidney Transplants: Insights From the MMDx Project. Transplantation. 2024 Jan 1;108(1):45-71. doi: 10.1097/TP.0000000000004624. Epub 2023 Dec 13. PMID 37310258
- [Result] Halloran PF, Reeve J, Madill-Thomsen KS, Kaur N, Ahmed E, Cantos C, Al Haj Baddar N, Demko Z, Liang N, Swenerton RK, Zimmermann BG, Van Hummelen P, Prewett A, Rabinowitz M, Tabriziani H, Gauthier P, Billings P; Trifecta Investigators*. Combining Donor-derived Cell-free DNA Fraction and Quantity to Detect Kidney Transplant Rejection Using Molecular Diagnoses and Histology as Confirmation. Transplantation. 2022 Dec 1;106(12):2435-2442. doi: 10.1097/TP.0000000000004212. Epub 2022 Nov 22. PMID 35765145
- [Result] Gauthier PT, Madill-Thomsen KS, Demko Z, Prewett A, Gauthier P, Halloran PF; Trifecta-Kidney Investigators. Distinct Molecular Processes Mediate Donor-derived Cell-free DNA Release From Kidney Transplants in Different Disease States. Transplantation. 2024 Apr 1;108(4):898-910. doi: 10.1097/TP.0000000000004877. Epub 2023 Dec 27. PMID 38150492
- [Result] Hidalgo LG, Madill-Thomsen KS, Reeve J, Mackova M, Gauthier P, Demko Z, Prewett A, Lee M, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Blosser CD, Bobba S, Brennan D, Bromberg J, Budde K, Chamienia A, Chow K, Ciszek M, Costa N, Deborska-Materkowska D, Debska-Slizien A, Domanski L, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Gryczman M, Gupta G, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kojc N, Konopa J, Kumar D, Lan J, Lowe D, Mazurkiewicz J, Miglinas M, Moinuddin I, Mueller T, Myslak M, Naumnik B, Paczek L, Patel A, Perkowska-Ptasinska A, Piecha G, Poggio E, Bloudickova SR, Regele H, Schachtner T, Shojai S, Sikosana MLN, Slatinska J, Smykal-Jankowiak K, Haler ZV, Viklicky O, Vucur K, Weir MR, Wiecek A, Zaky Z, Halloran PF. Improving the histologic detection of donor-specific antibody-negative antibody-mediated rejection in kidney transplants. Am J Transplant. 2025 Aug 23:S1600-6135(25)02943-0. doi: 10.1016/j.ajt.2025.08.029. Online ahead of print. PMID 40854490
- [Derived] Madill-Thomsen KS, Hidalgo LG, Demko ZP, Gauthier PM, Prewett A, Lowe D, Chang JJ, Mackova M, Budde K, Bromberg JS, Halloran PF; Trifecta-Kidney Study Group. Defining Relationships Among Tests for Kidney Transplant Antibody-Mediated Rejection. Kidney Int Rep. 2025 Jun 17;10(9):3225-3238. doi: 10.1016/j.ekir.2025.06.017. eCollection 2025 Sep. PMID 40980666
- [Derived] Halloran PF, Chang J, Mackova M, Madill-Thomsen KS, Akalin E, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Blosser CD, Bohmig G, Brennan D, Bromberg J, Budde K, Chamienia A, Chow K, Ciszek M, de Freitas D, Deborska-Materkowska D, Debska-Slizien A, Djamali A, Domanski L, Durlik M, Einecke G, Eskandary F, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Gryczman M, Gupta G, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kojc N, Konopa J, Lan J, Mannon RB, Matas A, Mazurkiewicz J, Miglinas M, Mueller T, Myslak M, Narins S, Naumnik B, Patel A, Perkowska-Ptasinska A, Picton M, Piecha G, Poggio E, Rajnochova Bloudickova S, Schachtner T, Shojai S, Sikosana ML, Slatinska J, Smykal-Jankowiak K, Solanki A, Veceric Haler Z, Viklicky O, Vucur K, Weir MR, Wiecek A, Wlodarczyk Z, Yang H, Zaky Z, Gauthier PT, Hinze C. A cross-sectional study of the role of epithelial cell injury in kidney transplant outcomes. JCI Insight. 2025 Apr 15;10(10):e188658. doi: 10.1172/jci.insight.188658. eCollection 2025 May 22. PMID 40232852
- [Derived] Halloran PF, Reeve J, Mackova M, Madill-Thomsen KS, Demko Z, Olymbios M, Campbell P, Melenovsky V, Gong T, Hall S, Stehlik J. Comparing Plasma Donor-derived Cell-free DNA to Gene Expression in Endomyocardial Biopsies in the Trifecta-Heart Study. Transplantation. 2024 Sep 1;108(9):1931-1942. doi: 10.1097/TP.0000000000004986. Epub 2024 Aug 20. PMID 38538559
- [Derived] Halloran PF, Madill-Thomsen KS. The Molecular Microscope Diagnostic System: Assessment of Rejection and Injury in Heart Transplant Biopsies. Transplantation. 2023 Jan 1;107(1):27-44. doi: 10.1097/TP.0000000000004323. Epub 2022 Dec 8. PMID 36508644